CLINICAL TRIAL: NCT01449760
Title: Ankle Sprain Rehabilitation With the Wii Balance Board
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Lara Allet, Principle investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09_116
Record Dates: First submitted 2011-10-05; First posted 2011-10-10 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Ankle Sprain
Keywords: Ankle sprain; Balance; Gait
MeSH Terms: conditions — Ankle Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No treatment (No Intervention)
- Physical Therapy (Active Comparator)
  Interventions: Other: Physical Therapy
- Wii Balance group (Experimental)
  Interventions: Other: Wii Balance Board

INTERVENTIONS:
Other: Physical Therapy — These patients have a standardized conventional therapy (i.e. 9 sessions of physical therapy over 6 weeks)
  Other Names: physiotherapy
  Arms: Physical Therapy
Other: Wii Balance Board — These patients get an instruction about how to install and use the Wii Balance Board ®. After the instruction they get the equipment for 6 weeks.
  Arms: Wii Balance group

SUMMARY:
Physical activity and in particular sport is beneficial to health. Nevertheless, some of these activities may create a risk of injury. Ankle sprain is the most common sport related injury. Sports that are causing the highest number of ankle sprains are: football (30%), handball-basketball-volleyball-rugby (24%), gymnastics sports (6%), skiing (6%), cycling (6%), athletics (4%) and contact sports (4%). A recent study in the Netherlands identified a total of 1.3 million sports injuries. 47% of these patients required medical care. The total costs (direct and indirect) were assessed 84.240.000 EUR per year.

Prospective studies demonstrated that athletes with a ankle sprain have a twofold risk of re-injury during the first year after the trauma, and in half of patients with an ankle sprain recurrence this could lead to instability or chronic pain of the ankle.

The Wii Balance Board ® is a tool that is increasingly used in the field of health. In some hospitals, therapists are beginning to use it for the rehabilitation of patients after surgery, fractures or strokes.

Patients are asked to complete their physical therapy session by practicing "sports" via video games such as skiing, bowling or hula hoop. Currently, there are no randomized controlled studies that publish on the effectiveness of this tool. Recently, a study investigated the efficacy of the Wii Balance Board ® to improve balance, strength, joint mobility and level of physical activity. After 10 weeks of training, people an increased strength and balance was found. However, these results still require statistical confirmation. Thus this objectives of this study are

* To assess the efficacy of exercise training with the Wii Balance Board ® Platform
* To evaluate the effectiveness of physical therapy (based on current guidelines)
* To compare these two types of care (conventional physiotherapy versus Wii) to a control group (non-treatment).

ELIGIBILITY:
Inclusion Criteria:

* Patients with an ankle sprain (grad 1 or 2), between 18 and 65 years old,

Exclusion Criteria:

* The subjects will not be included in the study if they are under 18 years
* They have other neurological or orthopedic disorders
* If taking medications (other than analgesics +/- NSAIDs prescribed during a sprain) that may influence the measurements.
* The patients with recurrent sprain of the ankle which was less than 12 months or who require surgery were also excluded.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2010-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in the balance performance(COP displacement in ML and AP direction) | 6 Weeks after the ankle sprain occured, after treatment (6 weeks) and in a 6 month follow up
  Change in the range of COP displacement during a single leg stance of 30 sec Change in the velocity of COP displacement during a single leg stance of 30 sec

SECONDARY OUTCOMES:
Change in several functional parameters | 6 weeks after ankle sprain, after treatment (6 weeks) and 6 month follow up
  * pain (VAS)
  * delay in return to work
  * delay in return to sport
  * passive joint mobility of the ankle in flexion and extension
  * isometric strength of the inverters and evertors, plantar and dorsal flexors
  * functional ankle instability evaluated with FAAM questionnaire
  * gait parameters (kinematics and electromyographic activity of peroneus, gastrocnemius and tibialis anterior)
  * performance during a forwrd jump "monopodal": distance and time to stabilize the ankle
  * incidence of recurrent sprains side: 12-month prospective follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Geneva, Geneva, Switzerland